CLINICAL TRIAL: NCT07049952
Title: BabyStrong II (Stimulating the Tragus for Neural Growth): A Randomized Controlled Trial of taVNS-Paired Bottle Feeding to Improve Oral Feeding
Brief Title: BabySTrong II taVNS Feeding Trial
Acronym: BabySTrong II
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Dorothea Jenkins, Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WCG 20250610; R42HD104409 (NIH)
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Feeding Delays; Neonates and Term Infants
Keywords: taVNS; feeding delays; infants; IDM; non-IDM; G-tube; transcutaneous auricular vagus nerve stimulation; Home NG feeds

STUDY DESIGN:
Intervention Model Description: We will stratify randomization based on non-IDM or IDM status (IDM is defined by obstetrical care providers, HgbA1C > 5.6%, or ketonuria), and then by oral feeding volume intake of <40ml/kg/d or >= 40ml/kg/d. For non-IDM we will use a device treatment: we will randomize 1:1 to active taVNS (Group T), or sham taVNS (Group C control non-IDM) paired with feeding twice daily for 14 days. For IDM cohort we will use a drug and device combination: we will randomize 1:1 to NAC and active taVNS-paired feeds (Group NT) or sham taVNS and placebo (Group C control IDM) for 14d. After the 14d period, all groups will receive 10d of open-label treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: parent
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Non-IDM active taVNS (Active Comparator): Non-IDM (Infants not product of diabetic mothers) will receive active taVNS with 2 feeds/day x 14 days
  Interventions: Device: taVNS
- Non-IDM Control (Sham Comparator): Non-IDM (Infants not product of diabetic mothers) will receive inactive/sham taVNS paired with 2 oral feedings a day for 14 days.
  Interventions: Device: inactive taVNS
- IDM NAC and active taVNS (Active Comparator): Infants of diabetic mothers will receive N-acetylcysteine by NG tube every 6h and active taVNS paired with 2 oral feedings a day, as a drug and device combination treatment for 14 days.
  Interventions: Combination Product: NAC and taVNS
- IDM Control (Sham Comparator): Infants of diabetic mothers will receive sterile water and inactive taVNS paired with 2 oral feedings a day, as a placebo drug and sham device combination treatment, for 14 days.
  Interventions: Combination Product: sterile water and inactive taVNS

INTERVENTIONS:
Device: taVNS — Active or inactive non-invasive vagus nerve stimulation of the auricular branch of the vagus nerve paired with 2 oral feedings/day for 14d
  Arms: Non-IDM active taVNS
Combination Product: NAC and taVNS — NAC 100 mg/kg diluted 1:3 with sterile water (or equal volume sterile water), q6h NG 1h before a feed for 4d prior to delivering active or sham taVNS paired with 2 feeds/day for 14d with NAC (or sterile water).
  Arms: IDM NAC and active taVNS
Device: inactive taVNS — inactive transcutaneous auricular vagus nerve stimulation with 2 feeds/day x 14 days
  Arms: Non-IDM Control
Combination Product: sterile water and inactive taVNS — Sterile water per NG tube every 6h for 4 days, then continuing with 14days of inactive taVNS paired with oral feeding
  Arms: IDM Control

SUMMARY:
The long-term goal of this project is to develop a therapy to assist pre-term and term infants with brain injury overcome difficulties in learning to feed so that infants may be discharged home with their families and avoid the burdens of of a gastrostomy tube (G-tube) or prolonged home nasogastric feeding. Few other therapies exist for infants who are not making progress with feeding volumes at term age.

To tackle this problem, we took the novel approach of pairing non-invasive nerve stimulation of the vagus nerve at the ear (taVNS) stimulation with the motor skills of feeding. In our pilot studies, 54% (19 out of 35) infants with feeding delays whose families were in discussions for G-tube placement, reached full oral feeds within 2 weeks, and infants who did not reach full feeds still improved their daily oral feeding volumes. Infants who got to full feeds showed stronger and more complex brain circuits associated with feeding motor skills.

With this trial we will test the BabySTrong taVNS feeding system in a multicenter, randomized, controlled, blinded trial to show how well this feeding system works in improving the daily feeding volumes, the days to full oral feeds, and/or the number of infants who avoid G-tube/ home NG placement, and increasing connections in brain circuits. If this groundbreaking new approach to infant feeding is successful, we may decrease how long infants are in the hospital, costs with Gtubes and home NG feeds, and family and care provider burdens. The findings from this proposal will be used in our FDA application for the BabySTrong feeding system.

DETAILED DESCRIPTION:
In this STTR, we will test the safety and efficacy of the BabyStrong taVNS feeding system in infants with feeding delays in a randomized, controlled, triple blinded, multicenter trial. With this safety and efficacy data, we intend to apply for FDA approval and commercially develop the BabyStrong feeding device.

Aim 1) Determine if twice daily active taVNS-paired feeding treatment increases the number of infants reaching full oral feeds or daily oral feeding volumes, or decreases the time to attain full oral feeds compared with infants receiving sham stimulation in a randomized, controlled, triple-blinded trial. We will randomize based on non-IDM or IDM status to 4 groups: IDMs will be randomized 1:1 to Active taVNS-paired feeds (Group T), or sham taVNS paired with feeds (Non-IDM Control); For IDM infants we will randomize 1:1 to N-acetylcysteine (NAC) and active taVNS-paired feeds (Group NT), or placebo and sham taVNS (IDM Control). Blinded randomized treatments will continue for 14 days, then all infants may progress to open label treatment, based on IDM status, for another 10days or less if full oral feeds or a decision to place a G-tube is reached. This study design will allow us to randomize to appropriate treatment based on IDM status. We will combine groups for analyses (Any active taVNS versus Control groups (IDM and Non-IDM combined), while controlling for IDM status. We hypothesize that any taVNS treatment (T + NT) will be effective at improving oral feeds over control (C).

We will also perform within stratified group analyses of active treatment versus control. We will use the non-IDM group results to support an FDA application.

Aim 2) Determine if active taVNS-paired feeding induces neuroplasticity compared with sham treated infants. We will measure diffusion kurtosis and tensor metrics in DKI scans at baseline and at the end of the 14d randomized treatment. We expect increased complexity (mean kurtosis) in corticospinal tracts in active vs sham groups.

Aim 3) Use safety and efficacy data to finalize an application for FDA approval of the BabyStrong, as a system with demonstrated potential to accelerate oromotor learning and decrease the need for Gubes and home NG feeds in infants.

ELIGIBILITY:
Inclusion Criteria:

* infants >39 weeks PMA making minimal progress in oral feeds
* trying to learn feeding for at least 2wks if beginning feeds at term (>37wks PMA), and 4wks if beginning feeds <36wks PMA,
* may po every feed without volume limitations by therapists

Exclusion Criteria:

* cardiomyopathy
* unstable apnea/bradycardia
* significant respiratory support (CPAP/ Vapotherm)
* unrepaired major congenital anomalies that affect safe po feeding or impose volume restrictions
* congenital syndromes unlikely to orally feed

Ages: 39 Weeks to 54 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2025-11-16 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
number of participants at full oral feeds | 24 days
  number of participants achieving full oral feeds receiving ANY active taVNS (groups T+NT), vs Control (IDM combined with Non IDM control groups), based on the randomized assignment.
rate of increase in daily oral feeding volumes | 7days / 10days
  mean daily rate of increase in oral feeding volumes in any active taVNS group (T+NT) vs Control (IDM and Non-IDM combined), based on randomized treatment assignment.

SECONDARY OUTCOMES:
time to full oral feeds | 24 days
  days to full oral feeds in any taVNS (groups T+NT) vs Control
Neuroplasticity via DKI | 14 days
  increased mean kurtosis (complexity ) or FA (integrity) in corticospinal tracts in any active taVNS (Groups T+ NT) vs Control groups

CONTACTS AND LOCATIONS:
Overall Officials: Dorothea D JENKINS, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Shawn Jenkins Children's Hospital, Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
We will preserve and share the subject level feeding, heart rate, and developmental test data with unique identifiers. The individual MRI scans will be preserved in Dicom and .rda format; and the VFSS in video files with same unique, coded identifiers.
Supporting Information: Study Protocol, ICF
Time Frame: data associated with a publication no later than the date of publication and all data at the end of the award and any NCE; DASH will control the end date for availability
Access Criteria: IPD will be placed in DASH, a controlled access data repository at NICHD. To request access of the data, researchers will use the standard processes, and the DASH Data Access Committee will decide which requests to grant.

REFERENCES:
- [Background] Badran BW, Dowdle LT, Mithoefer OJ, LaBate NT, Coatsworth J, Brown JC, DeVries WH, Austelle CW, McTeague LM, George MS. Neurophysiologic effects of transcutaneous auricular vagus nerve stimulation (taVNS) via electrical stimulation of the tragus: A concurrent taVNS/fMRI study and review. Brain Stimul. 2018 May-Jun;11(3):492-500. doi: 10.1016/j.brs.2017.12.009. Epub 2017 Dec 29. PMID 29361441
- [Background] Badran BW, Mithoefer OJ, Summer CE, LaBate NT, Glusman CE, Badran AW, DeVries WH, Summers PM, Austelle CW, McTeague LM, Borckardt JJ, George MS. Short trains of transcutaneous auricular vagus nerve stimulation (taVNS) have parameter-specific effects on heart rate. Brain Stimul. 2018 Jul-Aug;11(4):699-708. doi: 10.1016/j.brs.2018.04.004. Epub 2018 Apr 6. PMID 29716843
- [Background] Badran BW, Jenkins DD, DeVries WH, Dancy M, Summers PM, Mappin GM, Bernstein H, Bikson M, Coker-Bolt P, George MS. Transcutaneous auricular vagus nerve stimulation (taVNS) for improving oromotor function in newborns. Brain Stimul. 2018 Sep-Oct;11(5):1198-1200. doi: 10.1016/j.brs.2018.06.009. Epub 2018 Jun 30. No abstract available. PMID 30146041
- [Background] Moss HG, Brown TR, Wiest DB, Jenkins DD. N-Acetylcysteine rapidly replenishes central nervous system glutathione measured via magnetic resonance spectroscopy in human neonates with hypoxic-ischemic encephalopathy. J Cereb Blood Flow Metab. 2018 Jun;38(6):950-958. doi: 10.1177/0271678X18765828. Epub 2018 Mar 21. PMID 29561203
- [Background] Badran BW, Brown JC, Dowdle LT, Mithoefer OJ, LaBate NT, Coatsworth J, DeVries WH, Austelle CW, McTeague LM, Yu A, Bikson M, Jenkins DD, George MS. Tragus or cymba conchae? Investigating the anatomical foundation of transcutaneous auricular vagus nerve stimulation (taVNS). Brain Stimul. 2018 Jul-Aug;11(4):947-948. doi: 10.1016/j.brs.2018.06.003. Epub 2018 Jun 6. No abstract available. PMID 29895444
- [Background] Badran BW, Yu AB, Adair D, Mappin G, DeVries WH, Jenkins DD, George MS, Bikson M. Laboratory Administration of Transcutaneous Auricular Vagus Nerve Stimulation (taVNS): Technique, Targeting, and Considerations. J Vis Exp. 2019 Jan 7;(143):10.3791/58984. doi: 10.3791/58984. PMID 30663712
- [Background] Badran BW, Jenkins DD, Cook D, Thompson S, Dancy M, DeVries WH, Mappin G, Summers P, Bikson M, George MS. Transcutaneous Auricular Vagus Nerve Stimulation-Paired Rehabilitation for Oromotor Feeding Problems in Newborns: An Open-Label Pilot Study. Front Hum Neurosci. 2020 Mar 18;14:77. doi: 10.3389/fnhum.2020.00077. eCollection 2020. PMID 32256328
- [Background] Aljuhani T, Haskin H, Davis S, Reiner A, Moss HG, Badran BW, George MS, Jenkins D, Coker-Bolt P. Transcutaneous auricular vagus nerve stimulation (taVNS) given for poor feeding in at-risk infants also improves their motor abilities. J Pediatr Rehabil Med. 2022;15(3):447-457. doi: 10.3233/PRM-210090. PMID 36093716
- [Background] Jenkins DD, Moss HG, Adams LE, Hunt S, Dancy M, Huffman SM, Cook D, Jensen JH, Summers P, Thompson S, George MS, Badran BW. Higher Dose Noninvasive Transcutaneous Auricular Vagus Nerve Stimulation Increases Feeding Volumes and White Matter Microstructural Complexity in Open-Label Study of Infants Slated for Gastrostomy Tube. J Pediatr. 2023 Nov;262:113563. doi: 10.1016/j.jpeds.2023.113563. Epub 2023 Jun 16. PMID 37329979
- [Background] Aljuhani T, Coker-Bolt P, Katikaneni L, Ramakrishnan V, Brennan A, George MS, Badran BW, Jenkins D. Use of non-invasive transcutaneous auricular vagus nerve stimulation: neurodevelopmental and sensory follow-up. Front Hum Neurosci. 2023 Nov 9;17:1297325. doi: 10.3389/fnhum.2023.1297325. eCollection 2023. PMID 38021221
- [Background] Jenkins DD, Garner SS, Brennan A, Morris J, Bonham K, Adams L, Hunt S, Moss H, Badran BW, George MS, Wiest DB. Transcutaneous auricular vagus nerve stimulation may benefit from the addition of N-acetylcysteine to facilitate motor learning in infants of diabetic mothers failing oral feeds. Front Hum Neurosci. 2024 May 22;18:1373543. doi: 10.3389/fnhum.2024.1373543. eCollection 2024. PMID 38841121